CLINICAL TRIAL: NCT06812390
Title: Albumin Assisted Diuresis in Patients with Cirrhosis Decompensated by Ascites and Peripheral Edema, a Proof-of-concept Double Blind Randomized Trial
Brief Title: Albumin Assisted Diuresis in Patients with Cirrhosis and Ascites
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anahita Rabiee MD MHS (U.S. Federal Agency)
Collaborators: Grifols Shared Services North America Inc (Unknown)
Responsible Party: Sponsor-Investigator, Anahita Rabiee MD MHS, Staff Hepatologist, MD, MHS, VA Connecticut Healthcare System
Organization: VA Connecticut Healthcare System (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 1791319; 680800001061 (Other Grant/Funding Number: Grifols (Investigator initiated Sponsored Research))
Record Dates: First submitted 2025-02-01; First posted 2025-02-06 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Cirrhosis; Ascites Hepatic
Keywords: albumin; cirrhosis; ascites; diuresis
MeSH Terms: conditions — Fibrosis; Ascites | interventions — Albumins; Saline Solution

STUDY DESIGN:
Intervention Model Description: Proof of concept, randomized, cross over, double-blind placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Albumin first (Active Comparator): Albumin for one dose, followed by at least 14 day washout period, before crossing over to the alternate arm to receive placebo for one dose.
- Placebo first (Placebo Comparator): Placebo for one dose, followed by at least 14 day washout period, before crossing over to the alternate arm to receive albumin for one dose.
  Interventions: Drug: Albumin infusion (25% albumin); Drug: Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: Albumin infusion (25% albumin) — Albumin 25 gram infusion
  Arms: Placebo first
Drug: Normal Saline (0.9% NaCl) — 100 cc of normal saline
  Arms: Placebo first

SUMMARY:
A small, pilot proof-of-concept placebo-controlled trial to explore the effects of albumin on diuresis in patients with cirrhosis, ascites and lower extremity edema. We will additionally investigate albumin's effect on preventing neurohumoral activation, and acute kidney injury after diuresis.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient patients with decompensated cirrhosis with past or current ascites and persistent lower extremity edema despite oral diuretic titration
* Serum albumin of < 3.5 g/dL
* Age >=18 years old

Exclusion Criteria:

* Patients with GFR < 30mL/min/1.73 m2
* Changes in oral diuretic regimen in the past 7 days (**patients can enter the study after 7 days of the change)
* Large Volume paracentesis (LVP) in the past 7 days (**patients can enter the study after 7 days)
* Albumin infusion within the previous 14 days (** patients can enter the study after 14 days)
* Spontaneous Bacterial Peritonitis in the past month
* Active variceal bleeding
* Current Hepatic encephalopathy (>= Grade 2 based on West Haven criteria)
* Co-administration of other diuretics such as Hydrochlorothiazide (amiloride or eplerenone in place of spironolactone, and Bumex/Torsemide in place of furosemide are acceptable)
* Hypotension (Mean Arterial Pressure <65 mmHg, Systolic Blood pressure <90 mmHg)
* Severe hyponatremia (Sodium <125 mEq/L)
* previous diagnosis of overt heart failure (systolic EF < 50%)
* Baseline oxygen requirement
* Hypersensitivity to albumin preparations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in fractional excretion of sodium (FENa) | 6 hours (baseline vs hour 6 after albumin vs placebo administration)
  Change in fractional excretion of sodium (FENa) with administration of albumin vs placebo

SECONDARY OUTCOMES:
Changes in neuro hormonal markers | 6 hours and 24 hours
  Changes in neuro hormonal markers including norepinephrine, renin, aldosterone

CONTACTS AND LOCATIONS:
Locations (1):
- West Haven VA Medical Center, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No